CLINICAL TRIAL: NCT06895850
Title: Eccentric Cycling Vs. Standard Rehabilitation for Post-ICU Recovery in COVID-19 Survivors
Acronym: ECC-4-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Andres Bello (Other)
Responsible Party: Principal Investigator, Luis Penailillo, Head of the Exercise and Rehabilitation Science Lab, Universidad Nacional Andres Bello
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: COVID 19
Keywords: rehabilitation; hospitalization; eccentric cycling
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This study utilized a two-treatment crossover design. Each treatment was eight weeks in duration, with a two-week washout period. The order of treatments was randomized and counterbalanced.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants performed the eccentric cycling training for 8 weeks (experimental group)
  Interventions: Other: Eccentric cycling training
- Standard Rehabilitation (Active Comparator): The training protocol for STD REHAB consisted of the same 5 min warm-up protocol used in ECC, followed by three sets of 8 repetitions of bicep curls, triceps extensions, shoulder abduction, bodyweight squats, deadlifts, and leg abductions with an elastic band with 2 min inter-set rest. The resistance of the elastic band tension was progressively increased according to the participant's tolerance based on RPE. ECC training was programmed for ~20-30 min, while STD REHAB lasted ~60 min per session.
  Interventions: Other: Standar Rehabilitation

INTERVENTIONS:
Other: Eccentric cycling training — The training protocol for the ECC consisted of a 5-minute warm-up on a stationary ergometer (RS1 Go, Life fitness, USA) before completion of the prescribed workout. In the first two weeks, participants completed two sets of 10 minutes of eccentric cycling at an RPE between 9-11 with 2 minutes of inter-set rest. Then, during weeks 3-8, participants completed two sets of 15 min of eccentric cycling at an RPE between 13-15 with 2 min inter-set rest.
  Arms: Intervention
Other: Standar Rehabilitation — The training protocol for STD REHAB consisted of the same 5 min warm-up protocol used in ECC, followed by three sets of 8 repetitions of bicep curls, triceps extensions, shoulder abduction, bodyweight squats, deadlifts, and leg abductions with an elastic band with 2 min inter-set rest. The resistance of the elastic band tension was progressively increased according to the participant's tolerance based on RPE. ECC training was programmed for ~20-30 min, while STD REHAB lasted ~60 min per session.
  Arms: Standard Rehabilitation

SUMMARY:
We performed a longitudinal crossover clinical study on survivors of COVID-19. We compared a standard rehabilitation protocol using elastic bands versus a novel eccentric cycling training protocol in individuals who have been discharged after being hospitalized due to COVID-19. We assessed the effects of these two rehabilitation modalities on physical performance, quality of life, and cognitive function parameters. We found that both protocols induced significant improvements in all variables. However, eccentric cycling induced such improvements involving less time per session. These findings could significantly impact strategies to treat COVID-19 survivors, which is a novel and impactful contribution to the body of knowledge.

DETAILED DESCRIPTION:
Twenty patients (9 men, 11 women) between the ages of 30 and 60 years who had been hospitalized for COVID-19 in an ICU volunteered for this study. Participants were hospital-discharged at least 6 months before the start of the study and had not undergone rehabilitation after hospital discharge.

This study utilized a two-treatment crossover design. Each treatment was eight weeks in duration, with a two-week washout period. The order of treatments was randomized and counterbalanced. Twenty participants were recruited and completed this study. This sample was deemed sufficient as an a-priori power analysis (G*Power 3.1.9, Germany) estimated that 18 patients were required to test the anticipated effect, considering a statistical power of 0.8 and alpha <0.05. This effect was estimated based on the 18.7% increase in the 6-minute walking test observed after 12 weeks of eccentric training [10]. Considering a 10% dropout, we recruited 20 participants for this study.

Condition order was randomly arranged as either ECC then STD REHAB (n=10) or STD REHAB then ECC (n=10) to account for a potential order effect of treatments. Both interventions lasted eight weeks, and assessments were performed before and after the interventions. As shown in Fig. 1A, during the ECC participant performed eccentric cycling using an arm-and-leg motorized cycle ergometer (Model ABJ-107-2, Medical Technology Co LTD, China) while during the STD REHAB condition participants performed functional rehabilitation using strengthening exercises with elastic bands (Fig. 1B). During the 2-week wash-out period, the participants refrained from training in preparation for their second intervention.

2.3 Interventions The exercise intensity was matched between conditions throughout the intervention period using the 6-20 point rating of perceived exertion (RPE; Borg´s Scale) [10]. For both groups, RPE progressively increased during the first two weeks from 9 (very light) to 11 (fairly light), and then over the next five weeks from 13 (somewhat hard) to 15 (hard). Additionally, heart rate (HR) and blood pressure (Omron Serie 5/7156, USA), and oxygen saturation (Heal Force A3, CHOICEMMED, China) were measured immediately after all training sessions to quantify the cardiovascular demands of training, which were averaged between training sessions.

The training protocol for the ECC consisted of a 5-minute warm-up on a stationary ergometer (RS1 Go, Life fitness, USA) before completion of the prescribed workout. In the first two weeks, participants completed two sets of 10 minutes of eccentric cycling at an RPE between 9-11 with 2 minutes of inter-set rest. Then, during weeks 3-8, participants completed two sets of 15 min of eccentric cycling at an RPE between 13-15 with 2 min inter-set rest.

The training protocol for STD REHAB consisted of the same 5 min warm-up protocol used in ECC, followed by three sets of 8 repetitions of bicep curls, triceps extensions, shoulder abduction, bodyweight squats, deadlifts, and leg abductions with an elastic band with 2 min inter-set rest. The resistance of the elastic band tension was progressively increased according to the participant's tolerance based on RPE. ECC training was programmed for ~20-30 min, while STD REHAB lasted ~60 min per session.

ELIGIBILITY:
Inclusion Criteria:

* Participants were hospital-discharged at least 6 months before the start of the study and had not undergone rehabilitation after hospital discharge.

Exclusion Criteria:

* Patients who did not pass the medical check-up before the study (patients with myocarditis and/or abnormal troponins or electrocardiograms from the last three months), oxygen-dependent patients, those with musculoskeletal injuries, bedridden patients, disoriented patients, or those with severe mental disabilities were excluded due to being unsafe to exercise.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Muscle Strength (Medical Research Council; MRC) | Baseline, Pre- intervention (Eccentric cycling and Standard rehabilitation groups) and 8 week after interventions (post- Eccentric cycling and Standard rehabilitation groups)
  Manual strength of six muscle groups (shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, and ankle dorsiflexion) was evaluated bilaterally following the MRC scale guidelines [17]. Each muscle group was rated on a scale from 0 (paralysis) to 5 (normal strength). The MRC-sum score evaluates global muscle strength. The final score ranges from 0 (total paralysis) to 60 (normal muscle strength in all four limbs) [17].
Handgrip Strength | Baseline, Pre- intervention (Eccentric cycling and Standard rehabilitation groups) and 8 week after interventions (post- Eccentric cycling and Standard rehabilitation groups)
  Manual handgrip strength was evaluated with a hand dynamometer (Jamar, USA) with the participant, seated with the elbow at 90°, performing a maximum grip for 3 seconds, expressed in kilograms. Three attempts were made for the dominant upper limb, with a one-minute rest between attempts, and the highest of the three values was registered [18].
Six-Minute Walk Test (6MWT) | Baseline, Pre- intervention (Eccentric cycling and Standard rehabilitation groups) and 8 week after interventions (post- Eccentric cycling and Standard rehabilitation groups)
  The 6MWT measured the distance a person could walk in 6 minutes as quickly as possible [10]. It was conducted in a 30 m long corridor. If the participant experienced chest pain, dyspnoea, sweating, cyanosis, or chest discomfort during the test, the test was stopped, and the distance covered until the onset of symptoms was recorded.
One-Minute Sit-to-Stand Test | Baseline, Pre- intervention (Eccentric cycling and Standard rehabilitation groups) and 8 week after interventions (post- Eccentric cycling and Standard rehabilitation groups)
  The participants were asked to cross their arms with hands on the opposite shoulders and to sit and stand from the chair as many times as possible in one minute [19]. This test serves as an estimate of lower extremity power and functional capacity [19].
Timed up and go (TUG) | Baseline, Pre- intervention (Eccentric cycling and Standard rehabilitation groups) and 8 week after interventions (post- Eccentric cycling and Standard rehabilitation groups)
  Participants were instructed to rise from a chair, walk three meters, turn around a cone, walk back to the chair, and sit down with their back leaning against the backrest as quickly and safely as possible [10]. The time in seconds (s) needed to perform the entire sequence was recorded. Each participant performed the TUG in three attempts with a 2-minute rest between attempts, and the fastest time was used for further analyses.

SECONDARY OUTCOMES:
Body Composition | Baseline, Pre- intervention (Eccentric cycling and Standard rehabilitation groups) and 8 week after interventions (post- Eccentric cycling and Standard rehabilitation groups)
  Anthropometric measurements were taken between 8 and 10 am after an overnight fast, including weight (kg) and height (cm). Furthermore, multifrequency bioimpedanciometry (InBody 120, InBody Co., Ltd, Republic of Korea) was used to determine the whole-body fat and muscle mass percentage [15] before and after interventions.
Peak Expiratory Flow | Baseline, Pre- intervention (Eccentric cycling and Standard rehabilitation groups) and 8 week after interventions (post- Eccentric cycling and Standard rehabilitation groups)
  Pulmonary function was assessed with a mini-Wright peak flow meter (Clement Clarke, Mini-Wright PFM, United Kingdom) by measuring the maximum expiratory flow maintained for 10 milliseconds, expressed in L/min. This test was performed with the participant seated with their knees and hips flexed at 90°. In this position, participants performed a maximum inspiration, placed the device's mouthpiece in their mouth and sealed it with their lips and their nose clipped, and then was asked to breathe out as forcefully and quickly as possible. This manoeuvre was repeated thrice with a 2 min rest between each attempt, and the highest value achieved was recorded [16].
Post-COVID-19 Functional Status Scale (PCFS) | Baseline, Pre- intervention (Eccentric cycling and Standard rehabilitation groups) and 8 week after interventions (post- Eccentric cycling and Standard rehabilitation groups)
  The PCFS is a validated questionnaire to assess the functionality of COVID-19 survivors upon hospital discharge [20]. It consists of an interview with questions about daily living activities, instrumental activities, social activities, and lifestyle that the patient must rate from 0 (no limitations) to 4 (severe functional limitation).
Montreal Cognitive Assessment (MoCA) | Baseline, Pre- intervention (Eccentric cycling and Standard rehabilitation groups) and 8 week after interventions (post- Eccentric cycling and Standard rehabilitation groups)
  The MoCA test assesses cognitive function and takes approximately 10 minutes [22]. The MoCA evaluates orientation, short-term memory, visuospatial and executive functioning, language skills, abstraction, animal naming, and attention aspects through a guided questionnaire. The total score is a maximum of 30 points, with an additional point added if the person has no schooling. Scores below 26 points indicate cognitive dysfunction [22].
Barthel Index | Baseline, Pre- intervention (Eccentric cycling and Standard rehabilitation groups) and 8 week after interventions (post- Eccentric cycling and Standard rehabilitation groups)
  This instrument is widely used to assess a person's ability to perform basic activities of daily living, providing a quantitative estimate of the degree of dependence. Patients scored their capacity to perform ten activities encompassing personal hygiene, eating, and moving around the home. Each activity was scored from 0 to 5, with 0 being unable to do it and five being completely independent in performing the task. All items were summed, with scores of 0-20 classified as total dependence, 21-60 as severe dependence, 61-90 as moderate dependence, 91-99 as slight dependence, and 100 as completely independent [23].

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Andres Bello, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inostroza M, Valdes O, Tapia G, Nunez O, Kompen MJ, Nosaka K, Penailillo L. Effects of eccentric vs concentric cycling training on patients with moderate COPD. Eur J Appl Physiol. 2022 Feb;122(2):489-502. doi: 10.1007/s00421-021-04850-x. Epub 2021 Nov 20. PMID 34799753